CLINICAL TRIAL: NCT02162563
Title: Treatment Strategies in Colorectal Cancer Patients With Initially Unresectable Liver-only Metastases CAIRO5 a Randomized Phase 3 Study of the Dutch Colorectal Cancer Group (DCCG)
Brief Title: Treatment Strategies in Colorectal Cancer Patients With Initially Unresectable Liver-only Metastases
Acronym: CAIRO5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dutch Colorectal Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAIRO5; 2013-005435-24 (EudraCT Number)
Record Dates: First submitted 2014-06-05; First posted 2014-06-12 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: Colorectal cancer; Chemotherapy; Anti-EGFR; Liver metastases; R0 R1 liver resection; Resectability of liver; Liver expert panel
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol; Bevacizumab; Irinotecan; Leucovorin; Fluorouracil; Oxaliplatin; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm B: FOLFOXIRI & bevacizumab (inclusion completed) (Experimental): Patients with RAS or BRAF mutated and/or right-sided tumors will receive 5FU, irinotecan, oxaliplatin (FOLFOXIRI) and bevacizumab.
  Intervention: FOLFOXIRI with bevacizumab
  Interventions: Drug: FOLFOXIRI with bevacizumab
- Arm A: FOLFOX/FOLFIRI & bevacizumab (inclusion completed) (Active Comparator): Patients with RAS or BRAF mutated and/or right-sided tumors will receive doublet fluoropyrimidine-containing chemotherapy (FOLFOX or FOLFIRI), plus bevacizumab.
  Intervention: FOLFOX/FOLFIRI with bevacizumab
  Interventions: Drug: FOLFOX/ FOLFIRI with bevacizumab
- Arm D: FOLFOX/FOLFIRI & panitumumab (Experimental): Patients with RAS and BRAF wildtype and left-sided tumors will receive doublet fluoropyrimidine-containing chemotherapy (FOLFOX or FOLFIRI), plus panitumumab.
  Intervention: FOLFOX/FOLFIRI with panitumumab
  Interventions: Drug: FOLFOX/ FOLFIRI with panitumumab
- Arm C: FOLFOX/ FOLFIRI & bevacizumab (Active Comparator): Patients with RAS and BRAF wildtype and left-sided tumors will receive doublet fluoropyrimidine-containing chemotherapy (FOLFOX or FOLFIRI), plus bevacizumab.
  Intervention: FOLFOX/FOLFIRI with bevacizumab
  Interventions: Drug: FOLFOX/ FOLFIRI with bevacizumab

INTERVENTIONS:
Drug: FOLFOX/ FOLFIRI with bevacizumab — FOLFIRI + bevacizumab Bevacizumab 5 mg/kg in 15-30 minutes i.v., followed by irinotecan 180 mg/m2 i.v. in 60 minutes together with leucovorin 400 mg/m2 i.v. in 120 minutes, followed by bolus 5-fluorouracil 400 mg/m2 within 4 minutes, all on day 1, followed by continuous infusion of 5-fluorouracil 2400 mg/m2 in 46 hours, every 2 weeks
  FOLFOX6 + bevacizumab Bevacizumab 5 mg/kg in 15-30 minutes i.v., followed by oxaliplatin 85 mg/m2 i.v. together with leucovorin 400 mg/m2 i.v. in 120 minutes, followed by bolus 5FU 400 mg/m2 within 4 minutes, all on day 1, followed by continuous infusion of 5-fluorouracil 2400 mg/m2 in 46 hours, every 2 weeks
  Other Names: - bevacizumab; - irinotecan; - leucovorin; - 5-fluorouracil; - oxaliplatin
  Arms: Arm A: FOLFOX/FOLFIRI & bevacizumab (inclusion completed); Arm C: FOLFOX/ FOLFIRI & bevacizumab
Drug: FOLFOXIRI with bevacizumab — FOLFOXIRI + bevacizumab Bevacizumab 5 mg/kg in 15-30 minutes i.v., followed by irinotecan 165 mg/m2 i.v. in 60 minutes, followed by oxaliplatin 85 mg/m2 i.v. together with leucovorin 400 mg/m2 i.v. in 120 minutes, followed by continuous infusion of 5-fluorouracil 3200 mg/m2 in 46 hours, every 2 weeks
  Other Names: - bevacizumab; - irinotecan; - oxaliplatin; - leucovorin; - 5-fluorouracil
  Arms: Arm B: FOLFOXIRI & bevacizumab (inclusion completed)
Drug: FOLFOX/ FOLFIRI with panitumumab — FOLFIRI + panitumumab Panitumumab 6 mg/kg i.v. (1st dose in 60 minutes, if well tolerated subsequent doses in 30 minutes), followed by irinotecan 180 mg/m2 i.v. in 60 minutes together with leucovorin 400 mg/m2 i.v. in 120 minutes, followed by bolus 5-fluorouracil 400 mg/m2 within 4 minutes, all on day 1, followed by continuous infusion of 5-fluorouracil 2400 mg/m2 in 46 hours, every 2 weeks
  FOLFOX6 + panitumumab Panitumumab 6 mg/kg i.v. (1st dose in 60 minutes, if well tolerated subsequent doses in 30 minutes), followed by oxaliplatin 85 mg/m2 i.v. together with leucovorin 400 mg/m2 i.v. in 120 minutes, and bolus 5FU 400 mg/m2 within 4 minutes, all on day 1, followed by continuous infusion of 5-fluorouracil 2400 mg/m2 in 46 hours, every 2 weeks
  Other Names: - panitumumab; - irinotecan; - leucovorin; - 5-fluorouracil; - oxaliplatin
  Arms: Arm D: FOLFOX/FOLFIRI & panitumumab

SUMMARY:
Colorectal cancer patients with initially unresectable liver-only metastases may be cured after downsizing of metastases by neoadjuvant systemic therapy. However, the optimal neoadjuvant induction regimen has not been defined, and no consensus exist on criteria for resectability.

In this study colorectal cancer patients with initially unresectable liver-only metastases, as prospectively confirmed by an expert panel according to predefined criteria, will be tested for RAS and BRAF tumor mutation status and selected by location of primary tumor. Patients with RAS or BRAF mutant and/or right sided tumors will be randomised between doublet chemotherapy (FOLFOX or FOLFIRI) plus bevacizumab (schedule 1), and triple chemotherapy (FOLFOXIRI) plus bevacizumab (schedule 2). Patients with RAS AND BRAF wildtype AND left-sided primary tumors will be randomized between doublet chemotherapy (FOLFOX or FOLFIRI) plus either bevacizumab (schedule 1) or panitumumab (schedule 3). Patient imaging will be reviewed for resectability by a central panel, consisting of at least one radiologist and three surgeons every assessment. Central panel review will be performed prior to randomization as well as during treatment, as described in the protocol.

DETAILED DESCRIPTION:
Patients will be stratified for resectability of liver metastases (potentially resectable versus permanently unresectable), serum lactate dehydrogenase (LDH) (normal versus abnormal), BRAF mutation status (wildtype versus mutated), type of neoadjuvant chemotherapy (FOLFIRI versus FOLFOX) and hospital of registration.

Patients with RAS and BRAF wildtype and left-sided primary tumors will be randomised between FOLFOX or FOLFIRI plus either bevacizumab or panitumumab. The choice between FOLFOX or FOLFIRI is to the discretion of the local investigator, however, the treatment is restricted to regimens that are specified in the protocol. Patients with RAS or BRAF mutated and/or right-sided primary tumors will be randomized between FOLFOX/ FOLFIRI (investigator choice) plus bevacizumab or 5FU, irinotecan, oxaliplatin (FOLFOXIRI) plus bevacizumab.

Patients will be evaluated every 8 weeks by CT scan for disease status. The assigned systemic treatment should be continued for at least 6 months or earlier in case of resectability, progression of disease, unacceptable toxicity, or patient refusal. If after 6 months the panel concludes that the patient is still not resectable, it is highly unlikely that resectability will be achieved at all. Therefore the chemotherapy regimen may be reconsidered after 6 months of treatment. These patients should continue with the targeted drug in combination with chemotherapy, but the chemotherapy may be altered into a less toxic schedule such as fluoropyrimidine monotherapy. The targeted drug should be continued until progression or unacceptable toxicity. In patients who will become resectable and undergo secondary surgery of liver metastases, the total duration of preoperative and postoperative treatment together should be 6 months, with the chemotherapy schedule being administered according to the assigned treatment arm. However in these patients the targeted drug (bevacizumab or panitumumab) should not be continued after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of colorectal cancer
* Initially unresectable metastases confined to the liver according to CT scan, obtained ≤3 weeks prior to registration. Unresectability should be confirmed by the liver expertpanel. Patients with small (≤ 1 cm) extrahepatic lesions that are not clearly suspicious of metastases are eligible
* Known mutation status of RAS and BRAF
* WHO performance status 0-1 (Karnofsky performance status ≥ 70)
* Age ≥ 18 years
* No contraindications for liver surgery
* In case of primary tumor in situ: tumor should be resectable
* In case of resected primary tumor: adequate recovery from surgery
* Adequate organ functions, as determined by normal bone marrow function (Hb ≥ 6.0 mmol/L, absolute neutrophil count ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L), renal function (serum creatinine ≤ 1.5x ULN and creatinine clearance, Cockroft formula, ≥ 30 ml/min), liver function (serum bilirubin ≤ 2 x ULN, serum transaminases ≤ 5x ULN)
* Life expectancy > 12 weeks
* Expected adequacy of follow-up
* Written informed consent

Exclusion Criteria:

* Extrahepatic metastases, with the exception of small (≤ 1 cm) extrahepatic lesions that are not clearly suspicious of metastases
* Unresectable primary tumor
* Serious comorbidity or any other condition preventing the safe administration of study treatment (including both systemic treatment and surgery)
* Major cardiovascular events (myocardial infarction, severe/unstable angina, congestive heart failure, CVA) within 12 months before randomisation
* Uncontrolled hypertension, or unsatisfactory blood pressure control with ≥3 antihypertensive drugs
* Previous systemic treatment for metastatic disease; previous adjuvant treatment is allowed if completed ≥ 6 months prior to randomisation
* Previous surgery for metastatic disease
* Previous intolerance of study drugs in the adjuvant setting
* Pregnant or lactating women
* Second primary malignancy within the past 5 years with the exception of adequately treated in situ carcinoma of any organ or basal cell carcinoma of the skin, or second primary colorectal cancer.
* Any concomitant experimental treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2025-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2 years after last patient in study
  Time from registration until progression or death whichever comes first

SECONDARY OUTCOMES:
R0/1 secondary resection rate | 2 years after last patient in study
  R0/1 secondary resection rate in each of the 4 study arms upon neoadjuvant treatment with chemotherapy plus targeted therapy.
Median overall survival | 8 years after last patient in study
  From date of randomisation to death or last known to be alive
Response rate | 2 years after last patient in study
  Response according to RECIST 1.1
Toxicity (AE) | 2 years after last patient in study
  Patients will be evaluated for Adverse Events at the start of each treatment cycle according to CTCAE version 4.0.
Pathological complete response rate (pCR) | 2 years after last patient in study
  Pathological complete response rate (pCR) of the resected lesions
Postoperative morbidity | After surgery during two months
  Patients will be evaluated for surgical morbidity during 2 months. Postoperative morbidity will be scored according 'Clavien Dindo Grade'.
Correlation of evaluation by the panel with outcome | 2 years after last patient in study
  CT-scans will be reviewed for liver resectability by expert panel before randomisation and during neo-adjuvant treatment (every 8 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: C.J.A. Punt, Prof. dr., Principal Investigator — University Medical Center, Utrecht NL; R.J. Swijnenburg, Dr., Principal Investigator — Academic Medical Center, Amsterdam NL
Locations (56):
- Universitair ziekenhuis Antwerpen, Antwerp, Belgium
- Netherlands (55):
  - Flevoziekenhuis, Almere Stad, Flevoland
  - Gelre Ziekenhuis, Apeldoorn, Gelderland
  - Rijnstate ziekenhuis, Arnhem, Gelderland
  - Sint Jansdal Ziekenhuis, Harderwijk, Gelderland
  - Radboud UMC, Nijmegen, Gelderland
  - Streekziekenhuis Koningin Beatrix, Winterswijk, Gelderland
  - Atrium Medical Center, Heerlen, Limburg
  - Maastricht UMC+, Maastricht, Limburg
  - Laurentius Ziekenhuis, Roermond, Limburg
  - Orbis Medical Center, Sittard, Limburg
  - VieCuri Medisch Centrum, Venlo, Limburg
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant
  - Bravis Ziekenhuis, Bergen op Zoom, North Brabant
  - Amphia Ziekenhuis, Breda, North Brabant
  - Elkerliek Ziekenhuis, Helmond, North Brabant
  - Bravis Ziekenhuis, Roosendaal, North Brabant
  - Sint Elisabeth Ziekenhuis, Tilburg, North Brabant
  - TweeSteden Ziekenhuis, Tilburg, North Brabant
  - Bernhoven, Uden, North Brabant
  - Maxima Medisch Centrum, loc. Veldhoven, Veldhoven, North Brabant
  - Medisch Centrum Alkmaar, Alkmaar, North Holland
  - Amsterdam UMC, location AMC, Amsterdam, North Holland
  - Amsterdam UMC, location VUMC, Amsterdam, North Holland
  - Antoni van Leeuwenhoek, Amsterdam, North Holland
  - BovenIJ Ziekenhuis, Amsterdam, North Holland
  - OLVG, locatie Oost, Amsterdam, North Holland
  - OLVG, locatie West, Amsterdam, North Holland
  - Spaarne Gasthuis, Haarlem, North Holland
  - Tergooi, Hilversum, North Holland
  - Spaarne ziekenhuis, Hoofddorp, North Holland
  - Waterlandziekenhuis, Purmerend, North Holland
  - Zaans Medical Center, Zaandam, North Holland
  - Deventer Ziekenhuis, Deventer, Overijssel
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Ziekenhuisgroep Twente, Hengelo, Overijssel
  - Isala Klinieken, Zwolle, Overijssel
  - Ziekenhuis Nij Smellinghe, Drachten, Provincie Friesland
  - Medisch Centrum Leeuwarden, loc. Zuid, Leeuwarden, Provincie Friesland
  - Antonius Ziekenhuis, Sneek, Provincie Friesland
  - Martini Ziekenhuis, Groningen, Provincie Groningen
  - UMC Groningen, Groningen, Provincie Groningen
  - Reinier de Graaf, Delft, South Holland
  - Albert Schweitzer Ziekenhuis, Dordrecht, South Holland
  - LUMC, Leiden, South Holland
  - Erasmus MC, Rotterdam, South Holland
  - Ikazia Ziekenhuis, Rotterdam, South Holland
  - Maasstad Ziekenhuis, Rotterdam, South Holland
  - Sint Franciscus Gasthuis, Rotterdam, South Holland
  - Franciscus Vlietland, Schiedam, South Holland
  - Hagaziekenhuis, The Hague, South Holland
  - Medisch Centrum Haaglanden, Westeinde, The Hague, South Holland
  - UMC Utrecht, Utrecht, South Holland
  - Meander Medisch Centrum, Amersfoort, Utrecht
  - Sint Antonius Ziekenhuis, Nieuwegein, Utrecht
  - Admiraal de Ruyter ziekenhuis, Goes, Zeeland

IPD SHARING:
Plan to Share IPD: Yes
The data will be stored in the international ARCAD database which is available to other researchers.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: As of 2023
Access Criteria: Member of ARCAD

REFERENCES:
- [Derived] Bond MJG, Bolhuis K, Loosveld OJL, de Groot JWB, Droogendijk H, Helgason HH, Hendriks MP, Klaase JM, Kazemier G, Liem MSL, Rijken AM, Verhoef C, de Wilt JHW, de Jong KP, Gerhards MF, van Amerongen MJ, Engelbrecht MRW, van Lienden KP, Hermans JJ, Molenaar IQ, Grunhagen DJ, de Valk B, Haberkorn BCM, Kerver ED, Erdkamp F, van Alphen RJ, Mathijssen-van Stein D, Komurcu A, May AM, Swijnenburg RJ, Punt CJA; Dutch Colorectal Cancer Group. First-Line Systemic Treatment for Initially Unresectable Colorectal Liver Metastases: Post Hoc Analysis of the CAIRO5 Randomized Clinical Trial. JAMA Oncol. 2025 Jan 1;11(1):36-45. doi: 10.1001/jamaoncol.2024.5174. PMID 39570583
- [Derived] Wesdorp NJ, Zeeuw JM, Postma SCJ, Roor J, van Waesberghe JHTM, van den Bergh JE, Nota IM, Moos S, Kemna R, Vadakkumpadan F, Ambrozic C, van Dieren S, van Amerongen MJ, Chapelle T, Engelbrecht MRW, Gerhards MF, Grunhagen D, van Gulik TM, Hermans JJ, de Jong KP, Klaase JM, Liem MSL, van Lienden KP, Molenaar IQ, Patijn GA, Rijken AM, Ruers TM, Verhoef C, de Wilt JHW, Marquering HA, Stoker J, Swijnenburg RJ, Punt CJA, Huiskens J, Kazemier G. Deep learning models for automatic tumor segmentation and total tumor volume assessment in patients with colorectal liver metastases. Eur Radiol Exp. 2023 Dec 1;7(1):75. doi: 10.1186/s41747-023-00383-4. PMID 38038829
- [Derived] Bond MJG, Bolhuis K, Loosveld OJL, de Groot JWB, Droogendijk H, Helgason HH, Hendriks MP, Klaase JM, Kazemier G, Liem MSL, Rijken AM, Verhoef C, de Wilt JHW, de Jong KP, Gerhards MF, van Amerongen MJ, Engelbrecht MRW, van Lienden KP, Molenaar IQ, de Valk B, Haberkorn BCM, Kerver ED, Erdkamp F, van Alphen RJ, Mathijssen-van Stein D, Komurcu A, Lopez-Yurda M, Swijnenburg RJ, Punt CJA; Dutch Colorectal Cancer Study Group. First-line systemic treatment strategies in patients with initially unresectable colorectal cancer liver metastases (CAIRO5): an open-label, multicentre, randomised, controlled, phase 3 study from the Dutch Colorectal Cancer Group. Lancet Oncol. 2023 Jul;24(7):757-771. doi: 10.1016/S1470-2045(23)00219-X. Epub 2023 Jun 14. PMID 37329889
- [Derived] Wesdorp NJ, Kemna R, Bolhuis K, van Waesberghe JHTM, Nota IMGC, Struik F, Oulad Abdennabi I, Phoa SSKS, van Dieren S, van Amerongen MJ, Chapelle T, Dejong CHC, Engelbrecht MRW, Gerhards MF, Grunhagen D, van Gulik TM, Hermans JJ, de Jong KP, Klaase JM, Liem MSL, van Lienden KP, Molenaar IQ, Patijn GA, Rijken AM, Ruers TM, Verhoef C, de Wilt JHW, Swijnenburg RJ, Punt CJA, Huiskens J, Stoker J, Kazemier G; Dutch Colorectal Liver Expert Panel. Interobserver Variability in CT-based Morphologic Tumor Response Assessment of Colorectal Liver Metastases. Radiol Imaging Cancer. 2022 May;4(3):e210105. doi: 10.1148/rycan.210105. PMID 35522139
- [Derived] Huiskens J, van Gulik TM, van Lienden KP, Engelbrecht MR, Meijer GA, van Grieken NC, Schriek J, Keijser A, Mol L, Molenaar IQ, Verhoef C, de Jong KP, Dejong KH, Kazemier G, Ruers TM, de Wilt JH, van Tinteren H, Punt CJ. Treatment strategies in colorectal cancer patients with initially unresectable liver-only metastases, a study protocol of the randomised phase 3 CAIRO5 study of the Dutch Colorectal Cancer Group (DCCG). BMC Cancer. 2015 May 6;15:365. doi: 10.1186/s12885-015-1323-9. PMID 25943574
- See also: Website Dutch Colorectal Cancer Group — http://www.dccg.nl